CLINICAL TRIAL: NCT05594303
Title: Research on Chronic Obstructive Pulmonary Disease (COPD) Treatment by Transplantation of Autologous Bronchial Basal Cells
Brief Title: COPD Treatment by Transplantation of Autologous Bronchial Basal Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Regend Therapeutics (Industry)
Responsible Party: Principal Investigator, ShiYue Li, Professor, Guangzhou Institute of Respiratory Disease
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018001
Record Dates: First submitted 2019-03-26; First posted 2022-10-26 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; cell therapy; bronchial basal cells; autologous transplantation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronchial basal cells (Experimental): Treatment by autologous bronchial basal cells.
  Interventions: Biological: Autologuos transplantation of bronchial basal cells
- Control (No Intervention): No interventon.

INTERVENTIONS:
Biological: Autologuos transplantation of bronchial basal cells — Autologuos transplantation of bronchial basal cells
  Arms: Bronchial basal cells

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a group of disease characterized by obstructed airflow. Usually, the lung structure is gradually impaired along with the progression of the disease. Recently, the treatment of disease is challenged by shortage of approaches for regenerating the injured lung tissue. Here in this study, investigators intend to perform a single-centered, open, concurrent-controlled phase I/II clinical trial with autologous bronchial basal cells on COPD treatment since they were proved to regenerate lung tissue in animal models. The participants is recruited and divided into experiment group and control group. For patients from experiment group, bronchial basal cells will be isolated, expanded, carefully characterized in vitro and transplanted autologously into lung by fiberoptic bronchoscopy. No intervention is performed for patients from control group. During the study, the safety and efficacy will be evaluated on all the subjects by measuring the key indicators.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 40 to 75;
* Subjects diagnosed with COPD and meet the following standards: a. sustained airway obstruction; b. post-bronchodilator FEV1<80% predicted value;
* Subjects with DLCO<80% predicted value in spirometry;
* Subjects with a smoking history more than 10 pack-years (current smoker and former smoker);
* Subjects with stable condition for more than 4 weeks;
* Subjects tolerant to bronchoscopy;
* Subjects signed informed consent.

Exclusion Criteria:

* Pregnant or lactating women;
* Subjects with syphilis or any of HIV, HBV, HCV positive antibody;
* Subjects with any malignancy;
* Subjects requiring anti-infection (bacteria or virus) treatment by intravenous drugs;
* Subjects suffering from any of the following pulmonary diseases: asthma, active tuberculosis, pulmonary embolism, pneumothorax, pulmonary artery hypertension caused by other diseases;
* Subjects with a history of invasive or non-invasive mechanical ventilation in the past 4 weeks;
* Subjects suffering from other serious diseases, such as diabetes, myocardial infarction, unstable angina, cirrhosis, and acute glomerulonephritis;
* Subjects with leukopenia (WBC less than 4x10^9 / L) or agranulocytosis (WBC less than 1.5x10^9 / L or neutrophils less than 0.5x10^9 / L) caused by any reason;
* Subjects with severe renal impairment, serum creatinine> 1.5 times of the upper limit of normal;
* Subjects with liver disease or liver damage: ALT, AST, total bilirubin> 2 times of the upper limit of normal;
* Subjects with a history of mental illness or suicide risk, with a history of epilepsy or other central nervous system disorders;
* Subjects with severe arrhythmias (such as ventricular tachycardia, frequent superventricular tachycardia, atrial fibrillation, and atrial flutter, etc.) or cardiac degree II or above conduction abnormalities displayed via 12-lead ECG;
* Subjects with a history of alcohol or illicit drug abuse;
* Subjects allergic to products from cattle and pig;
* Subjects accepted by any other clinical trials within 3 months before the enrollment;
* Subjects with poor compliance, difficult to complete the study;
* Any other conditions that might increase the risk of subjects or interfere with the clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Diffusing capacity of the lung for carbon monoxide (DLCO) | Change from baseline DLCO at 3 months after transplantation
  It indicates the extent to which oxygen passes from the air sacs of the lungs into the blood

SECONDARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | Before transplantation, 3 months after transplantation, 6 months after transplantation and a year after transplantation
  It indicates the volume of air that can forcibly be blown out in first second, after full inspiration.
Forced vital capacity (FVC) | Before transplantation, 3 months after transplantation, 6 months after transplantation and a year after transplantation
  It indicates the volume of air that can forcibly be blown out after full inspiration.
The ratio of forced expiratory volume in one second to forced vital capacity (FEV1/FVC) | Before transplantation, 3 months after transplantation, 6 months after transplantation and a year after transplantation
  It represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration to the full vital capacity
Maximum voluntary ventilation (MVV) | Before transplantation, 3 months after transplantation, 6 months after transplantation and a year after transplantation
  It indicates the maximum amount of air that can be inhaled and exhaled within one minute
6-minute-walk test (6MWT) | Before transplantation, 3 months after transplantation, 6 months after transplantation and a year after transplantation
  An indicator to evaluate the exercise function of patients with moderate or severe pulmonary heart diseases.
Imaging of lung structure by computed tomography (CT) | Before transplantation, 3 months after transplantation, 6 months after transplantation and a year after transplantation
  Images of lung will be analyzed to indicate the newly-derived pulmonary structure.
Assess life quality affected by the respiratory problem by St. George's respiratory questionnaire (SGRQ) scale | Before transplantation, 3 months after transplantation, 6 months after transplantation and a year after transplantation
  Quality of life was assessed by St. George's respiratory questionnaire (SGRQ) scale. Total score, ranged from 0 to 100, is the sum of points from all items. A higher value represents a worse outcome.
Chronic obstructive pulmonary disease assessment test (CAT) | Before transplantation, 3 months after transplantation, 6 months after transplantation and a year after transplantation
  A patient-completed questionnaire assessing all aspects of the impact of Chronic obstructive pulmonary disease. Higher scores represent a worse outcome.
Diffusing capacity of the lung for carbon monoxide (DLCO) | Change from baseline DLCO at 6 months after transplantation
  It indicates the extent to which oxygen passes from the air sacs of the lungs into the blood
Diffusing capacity of the lung for carbon monoxide (DLCO) | Change from baseline DLCO at 12 months after transplantation
  It indicates the extent to which oxygen passes from the air sacs of the lungs into the blood

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, Principal Investigator — Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No